CLINICAL TRIAL: NCT01130987
Title: Implementing a Comprehensive Handoff Program to Improve Patient Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Walter Reed Army Medical Center (U.S. Federal Agency); Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christopher P. Landrigan, MD, MPH, Director, Sleep and Patient Safety Program, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2008P002191; BAA01 07005001
Record Dates: First submitted 2010-01-12; First posted 2010-05-26 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Medical Errors
Keywords: resident; intern; patient safety; medical error; time motion; handoff; sign-out; Resident Workflow; Resident Communications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Comprehensive Handoff Program (Experimental): Introduction of Computerized tool plus team training
  Interventions: Other: Computerized handoff tool; Behavioral: Team training

INTERVENTIONS:
Other: Computerized handoff tool — Computer program that facilitates accurate transmission of patient information between residents
Behavioral: Team training — Training in teamwork and reorganization of handoff processes to optimize transmission of information and team care

SUMMARY:
The investigators propose to test the hypothesis that implementation of a comprehensive handoff program (CHP) - i.e., implementation of a computerized handoff tool along with teamwork training for internal medicine residents on inpatient units at Walter Reed and Madigan Army Medical Centers - will lead to reductions in resident miscommunications / medical errors and improvements in workflow and experience on the wards.

DETAILED DESCRIPTION:
Following collection of baseline data on inpatient wards at both hospitals, teamwork training will be provided, accompanied by the introduction of a new computerized handoff tool that facilitates accurate transmission of data. The effects of this combined intervention on safety and workflow will be assessed on the intervention wards at both hospitals as compared with the historical control period.

ELIGIBILITY:
Inclusion Criteria:

* all internal medicine residents completing rotations through intervention units during data collection periods

Exclusion Criteria:

* none

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Rates of resident communication and total medical errors | July 2010

SECONDARY OUTCOMES:
Rates of all medical errors | July 2010
Rates of verbal miscommunications | July 2010
Rates of written miscommunications | July 2010
Resident workflow, especially time spent updating the signout; time spent at bedside; time spent at computer | July 2010
Resident care experience | July 2010

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Landrigan, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Walter Reed Army Medical Center, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Madigan Army Medical Center, Tacoma, Washington